CLINICAL TRIAL: NCT03865004
Title: Paracetamol Plus Morphine in ED
Brief Title: Combination Trial of Intravenous Paracetamol - Morphine for Treating Acute Renal Colic in Emergency Setting: An Optimum Treatment
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Akdeniz University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: firatbektas
Record Dates: First submitted 2019-03-04; First posted 2019-03-06 (Actual); Last update posted 2019-03-06 (Actual); Status verified 2019-03

CONDITIONS: Renal Colic
MeSH Terms: conditions — Renal Colic | interventions — dexketoprofen trometamol; Morphine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator)
  Interventions: Drug: Paracetamol+Morphine; Drug: Dexketoprofen plus Morphine; Drug: Placebo plus Morphine
- Paracetamol (Active Comparator)
  Interventions: Drug: Paracetamol+Morphine; Drug: Dexketoprofen plus Morphine; Drug: Placebo plus Morphine
- Dexketoprofene (Active Comparator)
  Interventions: Drug: Paracetamol+Morphine; Drug: Dexketoprofen plus Morphine; Drug: Placebo plus Morphine

INTERVENTIONS:
Drug: Paracetamol+Morphine — 1gr paracetamol plus 0.1 mg/kg morphine were performed simultanously
  Other Names: Parol
Drug: Dexketoprofen plus Morphine — Intravenous 75 mg Dexketoprofen plus 0,1 mg/kg morphine were performed simultanously
  Other Names: Arveles
Drug: Placebo plus Morphine — 100 cc NaCl plus 0.1 mg/kg morphine were performed simultanously
  Other Names: SF

SUMMARY:
This randomized, placebo-controlled trial evaluated the analgesic efficacy and safety of intravenous morphine-paracetamol combination and morphine-dexketoprofen combination morphine for the optimum treatment of renal colic. Combination of IV morphine and paracetamol is as effective and rapid as combination of IV Morphine and IV dexketoprophen for optimum treating of renal colic.

ELIGIBILITY:
Inclusion Criteria: Renal colic patients -

Exclusion Criteria: Not renal colic patients

-

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 136 (Actual)
Dates: Start 2015-10-17 (Actual); Primary Completion 2016-10-17 (Actual); Study Completion 2018-10-17 (Actual)

PRIMARY OUTCOMES:
pain reductions in VAS scores during the 60th and 90th minutes | 60 minutes

SECONDARY OUTCOMES:
Need for rescue analgesic | 30 minutes

IPD SHARING:
Plan to Share IPD: No